CLINICAL TRIAL: NCT03027804
Title: Database on Ross Operation Failures and Outcomes
Brief Title: Ross Operation Failure Database
Acronym: ROFDA
Status: Withdrawn | Type: Observational
Why Stopped: This study has been changed in systematic review and meta-analysis
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Golden Jubilee National Hospital (Other Government); University of Bern (Other); Pontifícia Universidade Católica do Paraná (Other); Ospedale San Donato (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CN-17-001
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Ross Operation; Pulmonary Autograft; Structural Valve Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ross Operation: Patients undergone Ross Operation. Patients requiring reoperation
  Interventions: Procedure: Ross Operation

INTERVENTIONS:
Procedure: Ross Operation — Replacement of the aortic valve by means of pulmonary artery autograft

SUMMARY:
A large multicentric registry to obtain data to analyse the pulmonary autograft (PA) failure phenomenon and feed more complex biomechanical models to be integrated with clinical imaging with the final aim to predict Ross operation's outcomes and define strategies to ameliorate its results.

DETAILED DESCRIPTION:
On the basis of the current knowledge on the outcomes of Ross Operation we aim to create a large multi centric registry in order to obtain data on the preoperative intraoperative management of these patients and on the postoperative long-term results of this procedure.

Patients data will be entered by the investigators in an electronic database Preoperative variables will include age, comorbidities, functional status, indications for surgery, morphology of the aortic valve Additional morphological data and aortic and pulmonary measurements will be taken intraoperatively Postoperative follow-up data including both clinical outcomes (mortality, reoperation for pulmonary autograft failure, major cardiac events, stroke, infection) and morphological measurements by means of CT scan or echocardiography, will be inserted.

Quality of life by means of SF12 and Minnesota living with heart failure questionnaire and EQ-5D score will be collected.

Follow-up endpoints are at discharge, 1 year 5 years 10 years 15 years and 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone (or undergoing) to Ross Operation

Exclusion Criteria:

* Patients requiring combined cardiac surgical procedure in association to Ross Operation

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergone (or undergoing) to Ross Operation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Survival | from inclusion to 20 years follow-up
  Death from any cause
Cardiac Death | from inclusion to 20 years follow-up
  Mortality due to cardiac cause
Reoperation for Pulmonary Autograft Failure | from inclusion to 20 years follow-up
  Need for reoperation due to failure of pulmonary autograft or valve degeneration
Stroke | from inclusion to 20 years follow-up
  neurological stroke with impairment
Rehospitalization for heart failure | from inclusion to 20 years follow-up
  Readmission to hospital for heart failure
Quality of life-1 | from inclusion to 20 years follow-up
  Quality of life as measured with SF-12
Quality of life-2 | from inclusion to 20 years follow-up
  Quality of life as measured with Minnesota living with heart failure questionnaire
Quality of life-3 | from inclusion to 20 years follow-up
  Quality of life as measured withEQ 5D score

SECONDARY OUTCOMES:
Postoperative complications | postoperative period (1-30 days)
  Combined outcome including bleeding, arrhythmia, respiratory failure, renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, MD, Principal Investigator — Centre Cardiologique du Nord
Locations (1):
- Centre Cardiologique Du Nord, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided